CLINICAL TRIAL: NCT04656509
Title: Effects of Short Duration High-intensity Interval Training on Peak Oxygen Consumption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-01-0132
Record Dates: First submitted 2020-10-12; First posted 2020-12-07 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-12

CONDITIONS: Cardiovascular Fitness
Keywords: exercise; cardiovascular fitness; sprinting; performance
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 4-s sprint inertial load training (Experimental): Participants trained three times a week for eight weeks following the training program consisting of 30 bouts of 4s all-out cycling on an inertial-load ergometer with progressively decreasing recovery time (30 to 24 to 15s).
  Interventions: Other: 4-s sprint inertial load training

INTERVENTIONS:
Other: 4-s sprint inertial load training — A program employing 30 bouts of 4s inertial load sprint training with progressively reduced recovery time (30 to 15 s) between sprints is effective for improving blood volume, VO2peak and maximal power.

SUMMARY:
High-intensity interval training (HIIT) is an effective tool to improve cardiovascular fitness and maximal anaerobic power. Different methods of HIIT have been studied but the effect of a maximal effort cycling and very short exercise time (i.e., 4-s) with short recovery time (15-30 s) and a high number of repetitions (i.e., 30 bouts) is unknown.

DETAILED DESCRIPTION:
The investigators examined the effects of training at maximal anaerobic power during cycling (PC) on maximal anaerobic power, peak oxygen consumption (VO2peak), and total blood volume in 11 young healthy individuals (age: 21.3±0.5 y) (6 men, 5 women). Methods: Participants trained three times a week for eight weeks performing a PC program consisting of 30 bouts of 4-s at an all-out intensity (i.e., 2 minutes of exercise per session). The cardiovascular stress progressively increased over the weeks by decreasing the recovery time between sprints (30 to 24 to 15-s) and thus session time decreased from 17 to < 10 min.

ELIGIBILITY:
Inclusion Criteria:

Young (18-30), Healthy, Recreationally active, but untrained (not meeting ACSM's recommendations of 150 min/week of moderate-vigorous aerobic exercise) -

Exclusion Criteria:

Cardiovascular disease Smoking Subjects who were exercising regularly (>75 min/week) were excluded.

-

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-04-24 (Actual)

PRIMARY OUTCOMES:
Cardiovascular changes | Pre and post training (8 weeks)
  Maximal oxygen consumption (VO2max) is an indicator of health and fitness. The investigators measured VO2max with a graded exercise using electronically braked cycling ergometer.
Blood volume changes | Pre and post training (8 weeks)
  Hematological variables can effect the performance of the people. The investigators measured total blood volume, red blood cell volume, and plasma volume before and after training.

SECONDARY OUTCOMES:
Performance changes | Pre and post training (8 weeks)
  Study participants trained at maximal anaerobic power for 4-s. Therefore, the investigators measured maximal anaerobic power with different testing methods.

CONTACTS AND LOCATIONS:
Overall Officials: Edward F Coyle, Ph.D., Study Director — University of Texas at Austin
Locations (1):
- Human Performance Laboratory, Department of Kinesiology and Health Education, the University of Texas at Austin, Austin, Texas, United States

REFERENCES:
- [Derived] Satiroglu R, Lalande S, Hong S, Nagel MJ, Coyle EF. Four-Second Power Cycling Training Increases Maximal Anaerobic Power, Peak Oxygen Consumption, and Total Blood Volume. Med Sci Sports Exerc. 2021 Dec 1;53(12):2536-2542. doi: 10.1249/MSS.0000000000002748. PMID 34310498